CLINICAL TRIAL: NCT06388694
Title: Pharmacist Management of Attention Deficit Hyperactivity Disorder Medication Refill Requests: A Randomized Clinical Trial
Brief Title: Pharmacist Management of Attention Deficit Hyperactivity Disorder Medication Refill Requests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RDO KPNC 24-056
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Attention-deficit Hyperactivity
MeSH Terms: interventions — Physicians, Primary Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist Care (Experimental): Pharmacists will provide ADHD medication refill orders in response to secure message requests by parents, under the authorization of appropriate physicians.
  Interventions: Other: Pharmacist Care
- Primary Care Physician Care (Active Comparator): Primary care pediatricians will provide ADHD medication refill orders in response to secure message requests by parents.
  Interventions: Other: Primary Care Physician Care

INTERVENTIONS:
Other: Pharmacist Care — Pharmacists will provide ADHD medication refill orders in response to secure message requests by parents, under the authorization of appropriate physicians.
  Arms: Pharmacist Care
Other: Primary Care Physician Care — Primary care pediatricians will provide ADHD medication refill orders in response to secure message requests by parents. This is usual care.
  Arms: Primary Care Physician Care

SUMMARY:
This cluster randomized trial will compare pharmacist management of secure message requests for refills of attention deficit hyperactivity medications with primary care physician management regarding quality of care, timeliness of service, and parent care experience.

DETAILED DESCRIPTION:
Importance. Enhancing the management of messages from patients and providing high-quality, consistent care are top priorities for The Permanente Medical Group (TPMG) and Kaiser Foundation Hospitals/Health Plan (KFH/P). A special extension of the Ryan Haight Act currently enables providers to prescribe controlled substances via telehealth interactions, but expires in December 2024. Information about the quality of care provided via telehealth prescribing of controlled substances by pharmacists and primary care physicians would be helpful to inform care delivery within Kaiser Permanente and beyond.

Objective. To compare pharmacist management of secure message requests for refills of attention deficit hyperactivity disorder (ADHD) medications with primary care physician management regarding quality of care, efficiency of service, and parent satisfaction.

Design, setting, and participants. This cluster randomized clinical trial will include parents of children in Kaiser Permanente Northern California who request ADHD medication refills via secure messages from April 29 to June 28, 2024. Of KPNC's 63 facilities eligible for inclusion, we will assign 32 to Pharmacist Care and 31 to PCP Care.

Intervention. In the intervention group, a regional team of pharmacists will manage ADHD medication refill requests made via secure message using a standard protocol. In the comparison group, primary care physicians (pediatricians and family medicine physicians) will manage these visits using a similar protocol.

Main Outcomes and Measures. The primary outcome is whether a patient who did not have a weight recorded in the 6 months before the refill request was referred for a primary care follow-up visit. Secondary outcomes are the days from the secure message request to the prescription order and medication fill, and parent satisfaction.

Potential Results. We will test the hypotheses that Pharmacist Care compared with PCP Care will have higher quality of care, faster time to prescriptions and fills, and higher patient satisfaction.

Potential Conclusions and Relevance. If pharmacist care for ADHD medication refill requests has better or similar outcomes compared with PCP care, this will provide evidence supporting continuation of this approach. This study's findings will be useful for KPNC and to inform discussions about renewing the special extension of the Ryan Haight Act that allows this approach.

ELIGIBILITY:
Inclusion Criteria:

* Parent or caregiver requested an ADHD medication refill via a secure message

Exclusion Criteria:

* The ADHD medication refill request was not straightforward and had to be handled by the primary care provider (and thus not eligible for random assignment to Pharmacist Care or PCP Care)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 315 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants appropriately referred for a follow-up weight check | within 7 days after the refill request
  Percentage of participants referred for a follow-up visit for a weight check, among those who had not had a weight check in the 6 months prior to the medication refill request

SECONDARY OUTCOMES:
Timeliness of care | within 14 days after the refill request
  Days between the refill request and the refill order, among patients eligible for a refill
Parent perception of effectiveness of care | within 3 weeks after the refill request
  Parent or caregiver perception of effectiveness of care given by the provider responding to the secure message request, as measured by a 5-point LIkert scale using Excellent, Very Good, Good, Fair, and Poor response options

CONTACTS AND LOCATIONS:
Overall Officials: Tracy A Lieu, Principal Investigator — Kaiser Permanente Northern California Division of Research
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lieu TA, Parry D, deLaunay A, Margaret Warton E, Prausnitz S, Ahmed O, Mancha MR, Smallberg E, Quesenberry C, Lee K, Reed M; Permanente Medical Group Virtual Care Study Team. Pharmacist care for attention-deficit/hyperactivity disorder electronic medication refills: A cluster randomized trial. J Manag Care Spec Pharm. 2025 Nov;31(11):1156-1165. doi: 10.18553/jmcp.2025.31.11.1156. PMID 41171067

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT06388694/Prot_SAP_000.pdf